CLINICAL TRIAL: NCT05404568
Title: The Hierarchical Rehabilitation After Total Knee Arthroplasty
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2022120
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-04

CONDITIONS: Rehabilitation；Arthroplasty, Replacement, Knee
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Total knee arthroplasty — We included patients with knee osteoarthritis who planned to take total knee arthroplasty

SUMMARY:
Knee osteoarthritis (KOA) is one of the diseases that seriously affect the quality of human life, resulting in a significant disease burden. Total knee arthroplasty (TKA) is one of the ultimate treatments for knee osteoarthritis. Functional recovery after total knee arthroplasty depends on rehabilitation. With the incidence rate of knee osteoarthritis increasing, the amount of knee replacement surgery is increasing rapidly, the demand for medical resources and medical expenditure has increased.

At present, there are many rehabilitation pathways after total knee arthroplasty, but there is no unified evidence-based medicine guide to guide postoperative rehabilitation. The current early rehabilitation pathways after total knee arthroplasty in China can be generally divided into three categories: inpatient rehabilitation, outpatient rehabilitation and home-based self-rehabilitation. The intensity and expenditure of rehabilitation treatment decrease in turn.

Individual differences among patients lead to different rehabilitation treatment needs for functional recovery. How to predict the rehabilitation needs of patients after total knee arthroplasty and choose an appropriate rehabilitation pathway based on themselves need to be solved.

We expected to establish a prediction model that we will be able to inform patients with knee osteoarthritis who just taken total knee arthroplasty and want to choose a pathway to rehabilitation by using the baseline status, that will help them to choose their best pathway to rehabilitation -- provide rehabilitation according to needs, save costs and improve the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* ① Knee osteoarthritis was diagnosed and total knee arthroplasty was planned;
* ② Good cognitive function, can cooperate and understand the contents of this test, and is willing to cooperate with rehabilitation evaluation and postoperative follow-up during perioperative period;
* ③ Aged 18 and above, voluntarily participated in the study and signed informed consent.

Exclusion Criteria:

* ① Accompanied by other local or systemic diseases that seriously affect the function of lower limbs, such as severe lumbar spinal stenosis, severe rheumatoid arthritis, etc;
* ② Patients have consciousness disorders, cognitive disorders, serious mental disorders and other diseases that affect limb function and cognition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with knee osteoarthritis who will take total knee arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Satisfaction of patients of total knee arthroplasty | 12 months after Total Knee Arthroplasty
  Satisfaction of patients（1-10 scoring）
HSS-KS score | 12 months after Total Knee Arthroplasty
  Hospital For Special Surgery Knee Score

SECONDARY OUTCOMES:
Visual analog scale of patients | 3 weeks，3 and 12 months after Total Knee Arthroplasty
  Visual analog scale of patients
Range of motion | 3 weeks，3 and 12 months after Total Knee Arthroplasty
  Range of motion of undergoing surgery
10mWT | 3 weeks，3 and 12 months after Total Knee Arthroplasty
  10 meters working test
WOMAC | 3 weeks，3 and 12 months after Total Knee Arthroplasty
  Western Ontario and McMaster Universities Osteoarthritis Index
SF-36 | 3 weeks，3 and 12 months after Total Knee Arthroplasty
  36-Item Short Form Survey
Satisfaction of patients of total knee arthroplasty | 3 weeks，3 months after Total Knee Arthroplasty
  Satisfaction of patients（1-10 scoring）
HSS-KS score | 3 weeks，3 months after Total Knee Arthroplasty
  Hospital For Special Surgery Knee Score

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No